CLINICAL TRIAL: NCT05683652
Title: The Effect of Education and Telephone Follow-up Given to Cancer Patients Receiving Immunotherapy on Symptom Management and Self-care Power
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Gamze ALINCAK, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: E-84892257-300-100327
Record Dates: First submitted 2022-06-21; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-06

CONDITIONS: Self Care; Symptom Management; Immunotherapy; Cancer Patient
Keywords: Immunotherapy; Symptom Management; Self care power

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TRAINING BOOKLET — Cancer patients in the intervention group, who will receive immunotherapy for the first time, will be given face-to-face training with the prepared training booklet and followed up by phone. Patients who received immunotherapy after the 1st, 2nd and 3rd cycles, respectively, will be called by phone. The researcher's phone number will be given to the intervention group patients and they will be told that they can call 24/7 if they experience any symptoms. The telephone interview form created by the researcher will be used during the monitoring by telephone.
  Other Names: Telephone follow up

SUMMARY:
This study, it was aimed to evaluate the effects of education and telephone follow-up given to cancer patients receiving immunotherapy on symptom management and self-care power. It is expected that the education given to the patients who will receive immunotherapy for the first time and the monitoring by phone, prevention of immunotherapy-related side effects, early recognition, and follow-up will reduce unnecessary hospital admissions and increase the self-care power of the patient.

DETAILED DESCRIPTION:
The research consists of two parts. For the qualitative part of the research; A semi-structured interview form was created. In this form, face-to-face interviews were conducted with the patients receiving immunotherapy about the symptoms they experienced, how they coped, and the subjects they wanted to learn.

Quantitative part for sample selection; G Power 3.1 statistical program was used to calculate the sample size of the study. After calculating the effect size as 0.73 by using the standard deviation and group averages of the Self-Care Scale of the study closest to the research, the sample calculation was made (Çetin,2020). According to this; The sample size was calculated with a total of 56 patients, 28 people in both groups, with a power of 85% in the 95% confidence interval. However, due to the possible losses in the number of patients, 33 people were planned for both groups, with a total of 66 patients (Çetin A.A.2020).

A randomization list created with a computer-based random number sequence was used to ensure the random distribution of the patients scheduled for immunotherapy to the groups (www.random.org). The patients were numbered according to the order of arrival, and the patients were assigned to the groups (intervention group with training and followed up by phone, and control group with routine follow-up) according to the numbers in the randomization list. Due to the nature of the study, the principal investigator and patients could not be blinded during grouping. However, single-blind randomization was achieved by blinding the evaluator groups.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in Turkish,
* Absence of any psychiatric disorder that will reduce the ability to comprehend and understand,
* Not having any physical discomfort in the area of hearing or speaking that would prevent telephone conversations,
* Will receive immunotherapy for the first time and only,
* Willingness to participate in the research,
* Willingness to participate in the research,
* Patients who agreed to participate in the study verbally and in writing were included in the study.

Exclusion Criteria:

* Not being voluntarily or willing to participate in the research,
* Will receive radiotherapy or chemotherapy together with immunotherapy,
* Not knowing that he will receive immunotherapy,
* Patients who did not accept to participate in the study were not included in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Nightingale Symptom Rating Scale | In patients receiving immunotherapy, the first measurements will be made at the end of the 1st cycle (the cycle is 28 days)
  Nightingale Symptom Assessment Scale (N-SDS) is a quality of life scale developed by Gülbeyaz Can and Adnan Aydıner in 2009 for cancer patients. Consisting of 38 items in total, the scale (N-CSS) has three sub-dimensions: Physical Well-Being (Physician) (items 1-4, 6-15, 23-27 and 37), Social Well-Being (SoIH) (5 and Articles 16-22) and Psychological Well-Being (PSYH) (Articles 28-36 and 38). When each item in the scale is used alone, it can be reflected how the cancer patients who are planned to receive or receiving chemotherapy are affected by the disease/treatment-related problems. In this Likert-type scale, the answer given by the patient to the evaluated item is scored as "0", if it is very little, "1", if it is a little, "2", if it is quite a lot, "3", and if it is too much, it is scored as "4". A high score indicates that the level of being affected by the disease/treatment-related problems is high.
Demographic and Medical Characteristics - Patient Information Form | It will meet within 3 months with patients who agree to participate in the study.
  It consists of a total of 8 questions created by the researcher after the literature review. 6 questions include medical characteristics, 2 questions include demographic characteristics.
Telephone Interview Form | Patients in the experimental group receiving immunotherapy will be followed up by phone for 3 months.
  atients who were given pre-immunotherapy training will be called after each cure and interviewed for symptom management. A telephone interview form was created by the researcher to record the interviews.
Phone Call Evaluation Form | It will be applied to the patients in the experimental group as a result of 3-month follow-up.
  A phone call evaluation form prepared by the researcher will be used to evaluate the phone calls made after each cure. It will be applied to the intervention group as a post-test.
Self Care Power Scale | The first measurements of the patients receiving immunotherapy will be done at the end of the 1st cycle (each cycle is 28 days)
  The scale used to measure an individual's self-care ability or self-care power was developed by Kearney and Fleicher (1979) in English with 43 items, and is a 35-item shortened Turkish form. The scale focused on individuals' self-assessment of their involvement in self-care actions. Each statement is scored from 0 to 4. Individuals' orientation towards self-care is determined by participants' responses on a 5-point Likert-type scale. Among the answer options, "Doesn't describe me at all" is given 0 points, the others are given 1 point for "Doesn't describe me very well", 2 points for "I have no idea", 3 points for "Describes me a little", and 4 points for "Describes me a lot".In the Turkishized scale, 8 items (3, 6, 9, 13, 19, 22, 26 and 31) are evaluated as negative and the scoring is reversed. The maximum score is 140. The high score obtained from the scale indicates the high level of self-care or self-care ability and power of the individual. There is no limit/cut off value.

SECONDARY OUTCOMES:
Nightingale Symptom Rating Scale | In patients receiving immunotherapy, the second measurements will be made at the end of the third cycle (the cycle is 28 days)
  Nightingale Symptom Assessment Scale (N-SDS) is a quality of life scale developed by Gülbeyaz Can and Adnan Aydıner in 2009 for cancer patients. Consisting of 38 items in total, the scale (N-CSS) has three sub-dimensions: Physical Well-Being (Physician) (items 1-4, 6-15, 23-27 and 37), Social Well-Being (SoIH) (5 and Articles 16-22) and Psychological Well-Being (PSYH) (Articles 28-36 and 38). When each item in the scale is used alone, it can be reflected how the cancer patients who are planned to receive or receiving chemotherapy are affected by the disease/treatment-related problems. In this Likert-type scale, the answer given by the patient to the evaluated item is scored as "0", if it is very little, "1", if it is a little, "2", if it is quite a lot, "3", and if it is too much, it is scored as "4". A high score indicates that the level of being affected by the disease/treatment-related problems is high.
Self Care Power Scale | n patients receiving immunotherapy, the second measurements will be made at the end of the third cycle (the cycle is 28 days)
  The scale used to measure an individual's self-care ability or self-care power was developed by Kearney and Fleicher (1979) in English with 43 items, and is a 35-item shortened Turkish form. The scale focused on individuals' self-assessment of their involvement in self-care actions. Each statement is scored from 0 to 4. Individuals' orientation towards self-care is determined by participants' responses on a 5-point Likert-type scale. Among the answer options, "Doesn't describe me at all" is given 0 points, the others are given 1 point for "Doesn't describe me very well", 2 points for "I have no idea", 3 points for "Describes me a little", and 4 points for "Describes me a lot".In the Turkishized scale, 8 items (3, 6, 9, 13, 19, 22, 26 and 31) are evaluated as negative and the scoring is reversed. The maximum score is 140. The high score obtained from the scale indicates the high level of self-care or self-care ability and power of the individual. There is no limit/cut off value.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided